CLINICAL TRIAL: NCT02294916
Title: Comparison of Pentax-AWS Airwayscope, Intubrite, AirTraq and Miller Laryngoscope for Tracheal Intubation by Nurses During Chest Compression in a Pediatric Manikin: A Randomised Crossover Trial.
Brief Title: Pediatric Intubation by Nurses
Acronym: NURS_ETI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/25
Record Dates: First submitted 2014-11-16; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Intubation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child ETI withoutchest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation without chest compressions.
  Interventions: Device: AWS; Device: Intubrite; Device: AirTraq; Device: MIL
- Child ETI with chest compressions (Experimental): Endotracheal intubation of mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: AWS; Device: Intubrite; Device: AirTraq; Device: MIL

INTERVENTIONS:
Device: AWS — Video-laryngoscopy 1
  Other Names: Pentax AWS
Device: Intubrite — Video-laryngoscopy 2
  Other Names: Intubrite Video Laryngoscope System VLS 6600
Device: AirTraq — Optical-laryngoscopy
  Other Names: AirTraq Optical Laryngoscope
Device: MIL — Direct-laryngoscopy
  Other Names: Miller Laryngoscope

SUMMARY:
The purpose of this study was to compare the Pentax AWS, Intubrite and AirTraq to Miller laryngoscope during pediatric resuscitation with and without chest compressions.

DETAILED DESCRIPTION:
Endotracheal intubation (ETI) is a life-saving procedure performed daily in emergency medicine. The European Resuscitation Council (ERC) 2010 cardiopulmonary resuscitation (CPR) guidelines suggest that intubators should be able to secure the airway without interrupting chest compression. However, ETI with uninterrupted chest compression in patients can be a very difficult skill to acquire.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel - nurses

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
VAS score | 1 day
  participants were asked which method they would prefer in a real-life resuscitation.
Cormack-Lehan scale | 1day
  self reported Cormack-Lehan scale during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland